CLINICAL TRIAL: NCT05787158
Title: Effects of Muscle Energy Techniques Versus Core Stability Exercises in Pelvic Girdle Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0546
Record Dates: First submitted 2023-03-15; First posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Pelvic Girdle Pain
MeSH Terms: conditions — Pelvic Girdle Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A: 20 patients were included in this group. This studygroup was assigned with basic treatment protocol with 15 minutes of TENS and thermal therapy for 10 minutes followed by muscle energy technique (Post facilitation stretching exercises). The intervention was given three days per weekfor six weeks. Each total session lasted for 45minutes. METs were applied for the weakened muscles.
  Interventions: Other: Muscle energy techniques
- Group B (Active Comparator): Group B: 20 Patients of this group were given core stability exercises by the female physical therapist in three different levels. Each level continued for a duration of two weeks in which the patients were trained for the exercises. The patients were provided sessions thrice per week with 2 sets of 10 repetitions and a hold of 10 second after TENS for 15 minutes and thermal therapy for 10 minutes.
  Interventions: Other: Muscle energy techniques

INTERVENTIONS:
Other: Muscle energy techniques — Group A: 20 patients were included in this group. This studygroup was assigned with basic treatment protocol with 15 minutes of TENS and thermal therapy for 10 minutes followed by muscle energy technique (Post facilitation stretching exercises). The intervention was given three days per weekfor six weeks. Each total session lasted for 45minutes. METs were applied for the weakened muscles. (21). Group B: 20 Patients of this group were given core stability exercises by the female physical therapist in three different levels. Each level continued for a duration of two weeks in which the patients were trained for the exercises. The patients were provided sessions thrice per week with 2 sets of 10 repetitions and a hold of 10 second after TENS for 15 minutes and thermal therapy for 10 minutes
  Other Names: core stability exercises

SUMMARY:
PGP is referred to as a specific form of LBP which occurs isolatedly as well as in combination with lumbar back pain. PGP localized to the anterior or posterior pelvis, most commonly located between the posterior iliac crest and gluteal folds especially around the SI joint. Pelvic girdle pain radiated to the posterior thigh

DETAILED DESCRIPTION:
Pelvic girdle pain (PGP) is known to be a musculoskeletal disorders which affects the pelvic bone. PGP is referred to as a specific form of LBP which occurs isolatedly as well as in combination with lumbar back pain. PGP localized to the anterior or posterior pelvis, most commonly located between the posterior iliac crest and gluteal folds especially around the SI joint. Pelvic girdle pain radiated to the posterior thigh. Moreover, it can also cause pain in the symphysis (1). Compared to lower back pain, PGP is substantially more painful and linked with functional limitations as standing, walking, sitting and changing positions are less tolerable in such patients (2). PGP is musculoskeletal in nature and is not caused by gynecological or urological conditions (3). Despite the fact that the cause of PGP is unknown, it is considered that it occurs due to many reasons such as trauma, arthritis, anatomical fault or it can be associated with pregnancy (4

ELIGIBILITY:
Inclusion Criteria:

* Females of 25 to 40 years were included in this study.(20)
* Female patients who gave birth at least 6 months before.(20)
* Females who gave birth through vaginal delivery.(20)
* Females with at least three positive pain provocative tests such as posterior pelvic pain provocation test (P4), active straight leg raise test (ASLR), thigh thrust, Patrick's Faber test, Gaenslen's test and distraction test.(20)
* History of pain around the pelvic girdle, lower back or between the posterior iliac crest and the gluteal fold, difficulty in walking and/or pain when putting weight on one leg

Exclusion Criteria:

* Females who suffered from grade 3 or 4 vaginal tears during their pregnancy (20)
* Females who underwent episiotomy during delivery (20)
* Females who delivered through caesarean section (20)
* Postpartum females with a history of trauma to the pelvic region (20)
* Postpartum females with a history of pelvic surgery
* Postpartum females with a history of other orthopedic disorders

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
VISUAL ANALOGUE SCALE | 12 weeks
  Visual Analogue scale is a numeric scale ranging from 1 to 10. These ranges show the intensity of pain where 1 shows no pain and 10 shows worst pain imaginations. It is a very reliable and valid tool with test-retest reliability of r = 0.96 and validity correlations of 0.86 to 0.95.
OSWESTRY DISABILITY INDEX | 12 weeks
  Oswestry Disability Index was calculated in order to find out the disability among patients. ODI evaluates disability related to Activities of Daily Living. This is considered to be the best tool for evaluating low back issues. It encompasses 10 questions with each question scoring five. Questions related to pain, personal care, walking, standing, lifting, sitting, sex life, sleeping, social life and travelling are included. The interpretation shows minimal disability if the patient score is 0-20%, moderate disability if the score is 20-40%, 40 - 60% severe disability, 60 - 80% crippled and 80 - 100 % depicting that the patient is either bed bound or overly expressing the symptoms
SF - 36 | 12 weeks
  This questionnaire is used to assess the functional performance in different domains of life like physical, body pain, mental, social and psychological. The questionnaire encompasses questions based on 7 domains of life. The minimum score of SF-36 is 0 which means that the functional performance is worst whereas the highest score is 100 which means that functional performance is best

CONTACTS AND LOCATIONS:
Overall Officials: Sobia Kanwal, tDpt, Principal Investigator — Riphah IU
Locations (1):
- Ghurki Trust Teaching Hospital., Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thabet AA, Alshehri MA. Efficacy of deep core stability exercise program in postpartum women with diastasis recti abdominis: a randomised controlled trial. J Musculoskelet Neuronal Interact. 2019 Mar 1;19(1):62-68. PMID 30839304
- [Background] Saleh MSM, Botla AMM, Elbehary NAM. Effect of core stability exercises on postpartum lumbopelvic pain: A randomized controlled trial. J Back Musculoskelet Rehabil. 2019;32(2):205-213. doi: 10.3233/BMR-181259. PMID 30282349
- [Background] Teymuri Z, Hosseinifar M, Sirousi M. The Effect of Stabilization Exercises on Pain, Disability, and Pelvic Floor Muscle Function in Postpartum Lumbopelvic Pain: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2018 Dec;97(12):885-891. doi: 10.1097/PHM.0000000000000993. PMID 29979205
- [Background] Almousa S, Lamprianidou E, Kitsoulis G. The effectiveness of stabilising exercises in pelvic girdle pain during pregnancy and after delivery: A systematic review. Physiother Res Int. 2018 Jan;23(1). doi: 10.1002/pri.1699. Epub 2017 Nov 8. PMID 29115735